CLINICAL TRIAL: NCT00857935
Title: A Pilot Study to Test the Operational Elements of an Actual Use Study Designed to Compare the Safety and Efficacy of NatrOVA Creme Rinse - 1% and NIX Creme Rinse in Subjects 6 Months of Age or Older With Pediculosis Capitis
Brief Title: A Safety and Efficacy Pilot Study Comparing NatrOVA Creme Rinse 1% and NIX Creme Rinse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ParaPRO LLC (Industry)
Responsible Party: Mark Moore, MD, Concentrics Research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPN-203-07; Concentrics 71007
Record Dates: First submitted 2009-03-05; First posted 2009-03-09 (Estimated); Last update posted 2009-03-09 (Estimated); Status verified 2009-03

CONDITIONS: Pediculosis Capitis; Head Lice
Keywords: Pediculosis Capitis; Head Lice
MeSH Terms: interventions — Permethrin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): NatrOVA Creme Rinse - 1%
  Interventions: Drug: NatrOVA Creme Rinse - 1%
- 2 (Active Comparator): NIX Creme Rinse
  Interventions: Drug: NIX Creme Rinse - 1% permethrin

INTERVENTIONS:
Drug: NatrOVA Creme Rinse - 1% — NatrOVA Creme Rinse, one or two, 10-minute topical treatments (7 days apart)
  Arms: 1
Drug: NIX Creme Rinse - 1% permethrin — NIX Creme Rinse: one or two, 10-minute topical treatments (7 days apart)
  Arms: 2

SUMMARY:
A pilot study to compare the safety and efficacy of NatrOVA Creme Rinse 1% to NIX Creme Rinse in subjects with Pediculosis Capitis

DETAILED DESCRIPTION:
A Phase 2b, randomized, single-site, investigator/evaluator blind, two-arm, parallel-group pilot study that tested the operational elements of an "Actual Use" study designed to evaluate the safety and efficacy of a 10-minute treatment and no-nit combing regimen of NatrOVA Creme Rinse 1% versus NIX Creme Rinse in subjects with at least a mild case of head lice.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 6 months of age or older
* Subject must have a head lice infestation present at baseline
* Subject/caregiver must read English or Spanish at a 7th grade level
* Subject must have an appropriately signed Informed Consent agreement
* Other members of the household with a lice infestation must be willing to be enrolled in the study or treat their infestations with a standard treatment
* Subject agreement to not use any other form of lice treatment during the course of the study
* Subject agreement to not cut or chemically treat their hair in the period between baseline and final, post-treatment visits

Exclusion Criteria:

* Individuals with a history of irritation or sensitivity to pediculicides or hair care products
* Individuals with any visible skin/scalp condition at the treatment site that could interfere with the evaluation
* Individuals previously treated with a pediculicide or any other head lice treatment product within 48 hours prior to enrollment
* Individuals receiving systemic or topical drugs that may interfere with the study results
* Individuals who have participated in a clinical trial within 30 days of enrollment
* Individuals with family members who are infested with lice but are unwilling or unable to enroll in the study or to use the standard course of lice treatment
* Females who are pregnant or nursing
* Sexually-active females not using effective contraception

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-03; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Efficacy of NatrOVA Creme Rinse-1% versus NIX Creme rinse, based on the presence or absence of live lice 14 days after the final treatment. | 14 days after last treatment

SECONDARY OUTCOMES:
Safety comparison between NatrOVA Creme Rinse-1% and NIX Creme Rinse, based on the occurrence of adverse events and any increase of scalp and/or ocular irritation, post-treatment. | 14 days after last treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mark Moore, MD, Principal Investigator — Concentrics Research
Locations (1):
- Concentrics Research, Indianapolis, Indiana, United States